CLINICAL TRIAL: NCT04146207
Title: SHR0302 and Prednisone As First Line Therapy for Chronic Graft Versus Host Disease Following Allogeneic Stem Cell Transplantation
Brief Title: SHR0302 and Steroid As First Line Therapy for Chronic GVHD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-cGVHD-2019002
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-01

CONDITIONS: Chronic GVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ivarmacitinib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- combination therapy (Experimental): Experimental: combination therapy There is only 1 arm. Combination therapy arm includes SHR0302 and Prednisone
  Prednisone 1mg/kg/d po，At the same time give SHR0302 QDpo；
  Interventions: Drug: SHR0302; Drug: Prednisone

INTERVENTIONS:
Drug: SHR0302 — SHR0302 po QD
Drug: Prednisone — Prednisone 1mg/kg/d po

SUMMARY:
The purpose of this study is to evaluate the efficacy of SHR0302 in combination with Prednisone as first line therapy in patients with moderate to severe chronic graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
Treatment: Once patients are diagnosed with chronic GVHD, the combination therapy should be initiated as soon as possible. 1. Prednisone: 1mg/kg/d po. Taper steroid every two weeks according to patient's response. 2. SHR0302 QD po. for at least 28 days. Indication for stopping SHR0302 treatment: 1. No response after SHR0302 treatment for 12 weeks. 2. Develop life-threatening complication. 3. ANC<0.5×10e9/L or PLT< 30×10e9/L.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old and ≤ 70 years old, male or female;
* Patients receiving allogeneic peripheral blood stem cell transplantation for hematological diseases;
* The primary hematological malignancies are completely relieved and are expected to be stable for at least 3 months;
* Chronic GVHD that was first attacked after transplantation and at least 100 days after transplantation, reached a moderate or severe level by NIH classification;
* There was no previous systemic treatment (including in vitro illumination [ECP]);
* The patient may be receiving other immunosuppressive agents to prevent or treat acute GVHD, but if the subject receives prednisone to prevent or treat acute GVHD, it must be <0.5 mg/kg/d or equivalent dose of other glucocorticoids;
* The chronic GVHD that has started hormone therapy does not exceed 72 hours;
* Karnofsky score > 60 points;
* Patients must be able to understand and are willing to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Can not tolerate prednisone dose 1mg / kg / d or equivalent dose of other glucocorticoids for the treatment of cGVHD;
* Receive any systemic treatment of cGVHD, except for corticosteroids that treat cGVHD within 72 hours prior to the signing of informed consent;
* Patients with GVHD overlap syndrome (NIH criteria);
* Treatment of acute GVHD has received other Jak inhibitors such as ruxolitinib;
* Pregnant or lactating women;
* The patient is judged by the investigator to have complications that may cause other risks;
* The patient is receiving other study medications;
* Patient blood routine: ANC <1.0 × 109 / L or PLT < 50 × 109 / L;
* Non-GVHD-related liver damage: the aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ratio is more than 3 times normal or the direct bilirubin normal value is more than 3 times;
* Renal dysfunction: endogenous creatinine clearance (Ccr) < 50mL/min or normal serum creatinine 1.5 times or more, regardless of hemodialysis treatment;
* Uncontrolled infections: hemodynamic instability associated with infection, or new signs or signs of infection, or new infections in imaging, persistent fever without symptoms or signs and cannot be ruled out Infected person
* People living with HIV;
* Active hepatitis B (HBV), active hepatitis C (HCV) requires antiviral therapy; patients with HBV activation risk refer to patients with hepatitis B surface antigen-positive or core antibody-positive patients who are not treated with anti-HBV;
* The patient's primary malignant disease recurs and the graft is rejected;
* Those who are allergic to known JAK inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SHR0302 and prednisone | After the first dose of SHR0302 or prednisone until 30 days after the last dose of SHR0302 or prednisone.
  The severity of adverse events is determined according to the CTCAE V5.0 criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) at week 4 | Within 4 weeks
  Response rate at week 4 (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014)
Overall response rate (ORR) at week 24 | Within 24 weeks
  Response rate at week 24 (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014)

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xianmin Song, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No